CLINICAL TRIAL: NCT03923010
Title: Itraconazole in the Management of Superficial Fungal Infections in India. A Pilot Study
Brief Title: A Study of Itraconazole in the Management of Superficial Fungal Infections in India
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Further recruitment not possible due to COVID 19 impact. Hence a decision to close study was taken by the sponsor in Aug 2020
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CR108518; R051211FUN4058 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-04-18; First posted 2019-04-22 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Mycoses
MeSH Terms: conditions — Mycoses | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Itraconazole (Experimental): Participants with Tinea cruris or Tinea corporis infection that have been prescribed itraconazole 200 milligram (mg) daily by their treating physician will be enrolled in this study. Participants will receive itraconazole 200 mg orally once daily for 7 days and at the discretion of the treating physician on Day 14. Participants will also get their regular clinical care at the discretion of their treating physician.
  Interventions: Drug: Itraconazole

INTERVENTIONS:
Drug: Itraconazole — Participants will receive itraconazole 200 mg orally once daily for 7 days and at the discretion of the treating physician on Day 14. Participants will also get their regular clinical care at the discretion of their treating physician.
  Other Names: JNJ-16269994

SUMMARY:
The purpose of this study is to estimate the proportion of participants prescribed itraconazole for Tinea cruris or Tinea corporis who have clinical response after 7 days of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with Tinea cruris or Tinea corporis with or without history of treatment
* Are prescribed itraconazole at 200 milligram/day orally for the treatment of T. cruris or T. corporis and taken once a day
* A woman of childbearing potential must have a negative highly sensitive serum (beta human chorionic gonadotropin [beta hCG]) at screening on Day -3 to 0 before start of study drug
* A woman must be (a) not of childbearing potential (b) of childbearing potential and: Practicing a highly effective method of contraception (failure rate of less than [<] 1 percentage [%] per year when used consistently and correctly) and agrees to remain on a highly effective method while receiving study drug and until 30 days after last dose (that is, the end of relevant systemic exposure)
* A male participant must wear a condom when engaging in any activity that allows for passage of ejaculate to another person. A male participant must agree not to donate sperm for the purpose of reproduction during the study and for a minimum 90 days after receiving the last dose of study drug

Exclusion Criteria:

* History of ventricular dysfunction such as congestive heart failure (CHF) or receiving treatment for CHF, liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances at any time prior to the start of study
* Known achlorhydria or on treatment of gastric acidity
* Presence of other dermatoses, example. psoriasis, seborrhoeic or atopic dermatitis
* Infected with organism with known or established resistance to itraconazole
* Co-existing fungal infection of other body area

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-27 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Clinical Response | Day 7 (End of Treatment)
  Percentage of participants with clinical response will be reported. Assessment of clinical response will be done by using Investigator Global Evaluation tool based on the signs and symptoms and clinical improvement scores. The percentage of clinical improvement will be measured at the score ranging from 1 to 5 where Score 1: Healed (absence of signs and symptoms), Score 2: Markedly improved (greater than [>] 50 percentage [%] clinical improvement), Score 3: Considerable residual lesion (less than [<] 50% clinical improvement), Score 4: No change (same as baseline), and Score 5: Worse (deterioration from baseline). Clinical response will be defined as having Scores 1 or 2 (healed or markedly improved).

SECONDARY OUTCOMES:
Percentage of Participants who Have Mycological Cure | Day 14
  Percentage of participants who have mycological cure will be reported. Mycological cure is defined as both culture and microscopy negative to causative fungi.
Plasma Concentrations of Itraconazole and Hydroxy-Itraconazole | Days 7 and 14: Pre-dose, 2 and 4.5 hours
  Plasma concentrations of itraconazole and hydroxy-itraconazole will be measured.
Baseline Minimum Inhibitory Concentration (MIC) of Itraconazole | Baseline (Day 0)
  Minimum inhibitory concentration of itraconazole toward fungal pathogens will be determined.
Percentage of Participants with Clinical Response | Day 14
  Percentage of participants with clinical response will be reported. Assessment of clinical response will be done by using Investigator Global Evaluation tool based on the signs and symptoms and clinical improvement scores. The percentage of clinical improvement will be measured at the score ranging from 1 to 5 where Score 1: Healed (Absence of signs and symptoms), Score 2: Markedly improved (greater than [>] 50 percentage [%] clinical improvement), Score 3: Considerable residual lesion (less than [<] 50% clinical improvement), Score 4: No change (same as baseline), and Score 5: Worse (deterioration from baseline). Clinical response will be defined as having Scores 1 or 2 (healed or markedly improved).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (4):
- India (4):
  - Post Graduate Institute of Medical Education & Research (PGIMER), Chandigarh
  - Sri Ramachandra Medical Centre, Chennai
  - Yenepoya Medical College, Mangalore
  - Lata Mangeshkar Hospital, Nagpur

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Handa S, Villasis-Keever A, Shenoy M, Anandan S, Bhrushundi M, Garodia N, Fife D, De Doncker P, Shalayda K, Hu P, Fonseca S, Cure-Bolt N. No evidence of resistance to itraconazole in a prospective real-world trial of dermatomycosis in India. PLoS One. 2023 Feb 14;18(2):e0281514. doi: 10.1371/journal.pone.0281514. eCollection 2023. PMID 36787305
- See also: Itraconazole in the Management of Superficial Fungal Infections in India. A Pilot Study — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR108518&attachmentIdentifier=6ff38044-aee3-45d2-80df-d52197752d2a&fileName=CR108518_CSR-Synopsis.pdf&versionIdentifier=